CLINICAL TRIAL: NCT01738035
Title: A Multicentre, Interventional Treatment, Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Two Different Doses of Nefecon in Primary IgA Nephropathy Patients at Risk of End-stage Renal Disease
Brief Title: The Effect of Nefecon® in Patients With Primary IgA Nephropathy at Risk of Developing End-stage Renal Disease
Acronym: NEFIGAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Calliditas Therapeutics AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nef-202; 2012-001923-11 (EudraCT Number)
Record Dates: First submitted 2012-07-25; First posted 2012-11-30 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Primary IgA Nephropathy
Keywords: IgA nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NEFECON 8 mg/day (Experimental): NEFECON 8 mg/day (2 active + 2 placebo capsules daily) for 9 months
  Interventions: Drug: NEFECON
- NEFECON 16 mg/day (Experimental): NEFECON 16 mg/day (4 active capsules daily) for 9 months
  Interventions: Drug: NEFECON
- Placebo (Placebo Comparator): Placebo (4 placebo capsules daily) for 9 months
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NEFECON — All patients will receive a maximum recommended daily dose of an ACEI and/or ARB (or maximum tolerated dose not exceeding the maximum recommended daily dose) for the duration of the treatment and follow-up phases.
  Other Names: Budesonide modified-released capsules (4 mg/capsule)
  Arms: NEFECON 16 mg/day; NEFECON 8 mg/day
Other: Placebo — All patients will receive a maximum recommended daily dose of an ACEI and/or ARB (or maximum tolerated dose not exceeding the maximum recommended daily dose) for the duration of the treatment and follow-up phases.
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate efficacy and safety of two different doses of NEFECON in the treatment of patients with primary IgA nephropathy (IgAN) at risk of developing end-stage renal disease, under rigorous blood pressure control with an angiotensin-converting enzyme inhibitor (ACEI) and/or angiotensin II receptor I blocker (ARB).

DETAILED DESCRIPTION:
NEFECON is an add-on treatment to other medications for nephropathy symptoms and kidney function, including ACEI and/or ARBs. Rigorous blood pressure control will be achieved over a 6-month Run-in Phase in which ACEI and/or ARB will be dosed to target a blood pressure of <130/80 mm Hg and UPCR <0.5 g/g. Patients who complete the Run-in Phase, and despite optimized ACEI and/or ARB therapy, have a UPCR ≥0.5 g/g OR urine protein ≥0.75 g/24hr will be eligible for randomization and entry into the treatment phase of the trial. Patients will remain on their ACEI and/or ARB dosing regimen for the duration of the trial.

Patients entering the treatment phase will be administered NEFECON (8 mg/day OR 16 mg/day) OR placebo for a phase of 9 months. A 3-month follow-up phase will follow on from the treatment phase, of which the first 2 weeks will be used to taper the dose of those patients that received 16 mg/day dosing to 8 mg/day, with the placebo and 8 mg/day groups receiving placebo to retain blinding.

ELIGIBILITY:
Screening Inclusion Criteria:

1. Female or male patients ≥18 years
2. Biopsy-verified IgA nephropathy
3. Urine protein creatinine ratio ≥0.5 g/g OR urine protein ≥0.75 g/24hr
4. Estimated GFR (using the CKD-EPI formula) OR measured GFR ≥50 mL/min per 1.73 m2 OR ≥45 mL/min per 1.73m2 for patients on a maximum recommended or maximum tolerated dose of an ACEI and/or ARB
5. Willing to change antihypertensive medication regimen if applicable
6. Willing and able to give informed consent

Screening Exclusion Criteria:

1. Secondary forms of IgA nephropathy as defined by the treating physician (for example, Henoch-Schönlein purpura patients and those with associated alcoholic cirrhosis)
2. Presence of crescent formation in ≥50% of glomeruli assessed on renal biopsy
3. Kidney transplanted patients 4. Severe gastrointestinal disorders (including peptic ulcer disease and inflammatory bowel disease) which may impair drug effect, or other conditions which could modify the effect of the trial drug as judged by the Investigator
4. Patients currently treated with systemic immunosuppressive or systemic corticosteroid drugs (excluding topical or nasal steroids) or have been previously treated for more than one week within the last 24 months.
5. Patients currently treated chronically (daily dosing) with inhaled corticosteroid drugs or have previously been treated chronically for more than one month within the last 12 months
6. Patients previously treated with immunosuppressive or systemic corticosteroids for the treatment of IgA nephropathy
7. Patients unable to take oral medication or intolerant to budesonide or other corticosteroid preparations
8. Patients with known allergy or intolerance to ACEI, ARB or to any component of the trial drug formulation
9. Patients with acute or chronic infectious disease incl. hepatitis, HIV positive patients and patients with chronic urinary tract infections
10. Severe liver disease according to the discretion of the Investigator
11. Patients with Type 1 or 2 diabetes
12. Patients with uncontrolled cardiovascular disease as judged by the Investigator
13. Patients with current malignancy or history of malignancy during the last three years
14. For women only; pregnant or breast feeding or unwilling to use adequate contraception during the trial (only women of child bearing potential)

Randomization Inclusion Criteria:

1. Completion of the Run-in Phase
2. Urine protein creatinine ratio ≥0.5 g/g OR urine protein ≥0.75 g/24hr
3. eGFR ≥45 mL/min per 1.73 m2 using CKD-EPI formula OR measured GFR ≥45 mL/min per 1.73 m2

Randomization Exclusion Criteria:

1. Unacceptable blood pressure defined as a systolic value >160 mm Hg or diastolic >100 mm Hg
2. eGFR (CKD-EPI) loss >30% over the entire duration of the Run-in Phase
3. For women only; pregnant or breast feeding or unwilling to use adequate contraception during the trial (only women of child bearing potential)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-12; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in urine protein creatinine ratio | 9 months

SECONDARY OUTCOMES:
Change from baseline in urine albumin creatinine ratio | 9 months
Change from baseline in 24 hour albuminuria | 9 months
Change from baseline in estimated GFR | 9 months

OTHER OUTCOMES:
Change from baseline in urine protein creatinine ratio | 3-12 months
Change in urine albumin creatinine ratio | 3-12 months
Change from baseline in 24 hour albuminuria | 3-12 months
Change from baseline in estimated GFR | 3-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Fellström, MD, PhD, Principal Investigator — Professor of Medicine Department of Medical Sciences, Renal Medicine Uppsala University Hospital, Sweden; Alex Mercer, PhD, Study Director — Pharmalink AB, Stockholm, Sweden
Locations (58):
- Belgium (5):
  - University Hospital of Antwerp, Antwerp
  - Imelda Hospital, Bonheiden
  - Ghent University Hospital, Ghent
  - University Hospitals Leuven, Leuven
  - Heilig Hartziekenhuis Roeselare-Menen, Roeselare
- Czechia (3):
  - University Hospital, Olomouc
  - Charles University & General University Hospital, Prague
  - Institut klinické a experimentální medicíny, Prague
- Denmark (3):
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense
- Finland (3):
  - Helsinki University Central Hospital, Helsinki
  - Tampere University Hospital, Tampere
  - Turku University Central Hospital, Turku
- Germany (18):
  - RWTH Aachen, Aachen
  - Klinikum Augsburg, Augsburg
  - Charité Hospital, Berlin
  - Charité-Virchow Clinic, Berlin
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Klinikum-Bremen-Mitte, Bremen
  - University Hospital Carl Gustav Carus, Dresden
  - Studienzentrum Karlstrasse, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsmedizin Göttingen, Göttingen
  - University Hospital, Heidelberg
  - University of Jena, Jena
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universität München, Munich
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Regensburg, Regensburg
  - Deutsche Klinik für Diagnostik, Wiesbaden
  - Würzburg University Hospital, Würzburg
- Italy (6):
  - Policlinico di Bari, Bari
  - Azienda Ospedaliera G. Brotzu, Cagliari
  - Ospedale A Manzoni, Lecco
  - Bassini Hospital, Milan
  - Ospedale S. G. Bosco, Torino
  - Belcolle Hospital, Viterbo
- University Medical Center, Leiden, Netherlands
- Spain (5):
  - Fundación Puigver, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - 12 de Octubre Hospital, Madrid
  - Fundación Jimenez Diaz Hospital, Madrid
  - Hospital Universitario Gregorio Marañon, Madrid
- Sweden (6):
  - Central sjukhuset, Karlstad
  - Karlstad Central Hospital, Karlstad
  - University Hospital, Linköping
  - Danderyds Hospital, Stockholm
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala
- United Kingdom (8):
  - Belfast City Hospital, Belfast
  - Ulster Hospital, Belfast
  - Royal Derby Hospital, Derby
  - Edinburgh Royal Infirmary, Edinburgh
  - Western Infirmary, Glasgow
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - Leicester General Hospital, Leicester
  - James Cook University Hospital, Middlesbrough

REFERENCES:
- [Derived] Fellstrom BC, Barratt J, Cook H, Coppo R, Feehally J, de Fijter JW, Floege J, Hetzel G, Jardine AG, Locatelli F, Maes BD, Mercer A, Ortiz F, Praga M, Sorensen SS, Tesar V, Del Vecchio L; NEFIGAN Trial Investigators. Targeted-release budesonide versus placebo in patients with IgA nephropathy (NEFIGAN): a double-blind, randomised, placebo-controlled phase 2b trial. Lancet. 2017 May 27;389(10084):2117-2127. doi: 10.1016/S0140-6736(17)30550-0. Epub 2017 Mar 28. PMID 28363480
- [Derived] Yeo SC, Liew A, Barratt J. Emerging therapies in immunoglobulin A nephropathy. Nephrology (Carlton). 2015 Nov;20(11):788-800. doi: 10.1111/nep.12527. PMID 26032537